CLINICAL TRIAL: NCT06298721
Title: Improving Total Knee Arthroplasty Dissatisfaction at 1-year Through a Personalized Approach Focusing on PROMs Phenotypes: A Randomized Controlled Trial
Brief Title: Improving Total Knee Arthroplasty Dissatisfaction Through a Personalized Approach Focusing on PROMs Phenotypes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Association of Hip and Knee Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-885
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis; Knee Arthropathy; Surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care TKA (Active Comparator): Patients scheduled to undergo TKA at Cleveland Clinic will follow the standardized TKA Care Pathway as part of Standard of care. Patients enter the TKA care path after consenting to undergo TKA for symptomatic knee pain that has not relieved with nonoperative measures. They stay in the care path until 90-days after the operation is complete. The TKA care path guides the care delivered through the preoperative, intraoperative and postoperative phases.
  Interventions: Behavioral: Standard of Care TKA
- Standard of Care TKA + Personalized Outcome Prediction Tool with targeted interventions (Experimental): Patients who are identified to have a TKA PROMs phenotype which includes lower than median scores for VR-12 MCS will be further screened for:
  Distress ➔ using the NCCN Distress Thermometer (DT) Depression ➔ using the Patient Health Questionnaire-9 Those patients with a score ≥ 8 on the DT, or a score ≥ 10 on the PHQ-9, or any response other than 0 to question 9 on the PHQ-9 will have a consult with Psychiatry and Behavioral Science to determine a mental health diagnosis.
  Patients who are identified to have a TKA PROMS phenotype which includes lower than median scores for KOOS-PS (score of =<51.5) will be scheduled for a 4 to 8 week intervention of pre-rehabilitation. All patients who undergo the PT intervention will have a an assessment before and after the rehab TKA.
  Interventions: Behavioral: Personalized outcome prediction tool + targeted interventions

INTERVENTIONS:
Behavioral: Personalized outcome prediction tool + targeted interventions — * TKA Personalized Outcome Prediction Tool to aid in setting expectations
  * Mental Health Screening/Intervention
  * Physical Therapy Pre-surgery Assessments & Rehabilitation
  Arms: Standard of Care TKA + Personalized Outcome Prediction Tool with targeted interventions
Behavioral: Standard of Care TKA — - Standard of care preoperative TKA clinic appointment to discuss plan for surgery and get consent
  Arms: Standard of Care TKA

SUMMARY:
This study is a randomized controlled trial to assess whether the implementation of a TKA Personalized Outcome Prediction Tool to set expectation, in addition to targeted interventions to address patients with poor baseline mental health and poor physical function, improves satisfaction at 1-year (when compared to standard of care).

DETAILED DESCRIPTION:
The potential candidates for the study are patients scheduled for primary TKA. Scheduled patients will be sent an invitation letter detailing the study's objectives and design. Should they choose to take part, individuals will be requested to utilize MyChart for the completion of PROMs. The information gathered from these PROMs will play a pivotal role in assessing their suitability for inclusion in the study. Subsequently, once deemed eligible, our coordinator will arrange a convenient session to meticulously review and facilitate the signing of the informed consent form (enrollment visit). This enrollment visit will take place approximately 2-3 months prior to the scheduled surgery. Subsequently, enrolled patients will be randomized in a 1:1 ratio to:

i) Standard of Care ii) Standard of Care + TKA Personalized Outcome Prediction Tool (Mental Health Screening/Intervention & Physical Therapy Pre-surgery Assessments/Intervention)

TKA Personalized Outcome Prediction Tool aids in setting expectations for surgery and the results (calculated from patient information and baseline PROMs) will be provided and discussed with the patients by the surgeon.

The primary outcome of the study will be the proportion of patients who fail treatment, defined as patients who answer "no" to the PASS anchor question at 1-year postoperative. The treatment and control groups will be compared using a chi-square test between the randomized groups with p=0.05 as the threshold for statistical significance. We will follow the intent-to-treat principle, and patients assigned to the treatment/intervention arm will be analyzed as such regardless of his/her compliance with the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject (Age >18 and < 80 years of age)
2. The subject is proficient in the English language
3. The patient is voluntarily prepared to sign the 'Informed Consent Form'
4. The patient is scheduled for a unilateral primary TKA
5. TKA PROMs Phenotypes with higher risk of dissatisfaction
6. Patient is willing and able to complete the protocol required follow-up

Exclusion Criteria:

1. Patient requires simultaneous or staged bilateral knee replacements, staged <90 days apart
2. Patients undergoing revision TKA
3. Inflammatory arthritis
4. History of infection in the joint undergoing TKA
5. Patient is considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Satisfaction at 1 year | 1 year
  Patient Acceptable Symptom State (PASS) anchoring question of: "Taking into account all the activity you have during your daily life, your level of pain and also your activity limitations and participation restrictions, do you consider the current state of your knee satisfactory?" to measure satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas S Piuzzi, MD, Principal Investigator — Cleveland Clinic Ohio
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No